CLINICAL TRIAL: NCT00415311
Title: A Multicenter, Open-Label, Randomized, Phase 1B Study Evaluating the Safety and Tolerability of Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) in Liver Transplant Recipients
Brief Title: A Multicenter Study Evaluating the Safety and Tolerability of Intravenous rhMBL in Liver Transplant Recipients.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Nazish Huq, Clinical Project Manager, Enzon Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2232-02
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; rhMBL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0 mg/kg (Other)
  Interventions: Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL)
- 0.5 mg/kg (Other)
  Interventions: Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL)
- 1.0 mg/kg (Other)
  Interventions: Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL)

INTERVENTIONS:
Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) — Intravenous(i.v.) administration for 8 weeks. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 0 mg/kg
Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) — Intravenous(i.v.) administration for 8 weeks. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 0.5 mg/kg
Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) — Intravenous(i.v.) administration for 8 weeks. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 1.0 mg/kg

SUMMARY:
This is a multicenter, open-label, randomized, Phase 1B study evaluating liver transplant recipients receiving rhMBL (2 cohorts) or without rhMBL (1 cohort).

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, Phase 1B study evaluating liver transplant recipients receiving rhMBL (2 cohorts) or without rhMBL (1 cohort).

Patients will have received an orthotopic liver transplant (OLT) or a living related donor (LRD) liver transplant. Patients in all cohorts are to receive immunosuppressant therapy and anti-infectious prophylactic supportive therapy according to institutional standards.

The donor's mannose-binding lectin (MBL) genotype will be evaluated to determine the liver transplant recipient's study eligibility. For recipients receiving an OLT, a sample of liver tissue or lymph nodes will be collected from the donor liver at the time of organ harvest for MBL genotyping. For recipients receiving a LRD transplant, the MBL genotype of the LRD will be determined in a companion protocol, "Screening Protocol to Evaluate Mannose-Binding Lectin (MBL) Genotype in Living Related Donors for Liver Transplant Recipients." A recipient whose donor has an A/O or O/O MBL genotype will be eligible to participate in this study.

Patients will be randomized in a 2:2:1 ratio to receive up to 8 intravenous (i.v.) infusions of rhMBL at a dose of 0.5 or 1.0 mg/kg, or to receive no rhMBL, respectively. Approximately 20 patients will be treated in each of the 2 rhMBL arms, and approximately 10 patients will be treated with standard immunosuppressive agents and anti-infectious prophylaxis but not with rhMBL.

Cohort 1

* Number of Patients 20
* rhMBL (mg/kg) 0.5

Cohort 2

* Number of Patients 20
* rhMBL (mg/kg) 1.0

Cohort 3

* Number of Patients 10
* rhMBL (mg/kg) None

ELIGIBILITY:
Major Inclusion Criteria: Patients must meet all of the following criteria to be eligible for enrollment into the study:

* Capable of understanding the protocol requirements and risks and providing written informed consent.
* Scheduled to undergo OLT or LRD liver transplantation (single organ). Split grafts will not be allowed from OLT donors.
* Donor has an MBL genotype of A/O or O/O.
* Age ≥18 years old.
* Willing to receive transfusions of blood products.

Any patient who has given informed consent to participate in the clinical study and who meets all entry criteria for the study may participate in the genetic part of the study.

Exclusion Criteria: Patients meeting any of the following exclusion criteria will not be eligible for enrollment.

* Concurrent serious medical illness, in the judgment of the principal investigator (PI), which could potentially interfere with protocol compliance.
* Positive screening pregnancy test or is breast-feeding.
* Female or male patient of reproductive capacity unwilling to use methods appropriate to prevent pregnancy during this study.
* Any condition that, in the opinion of the PI or Enzon makes the patient unsuitable for the study.
* Current participation in another clinical study with an investigational agent and/or use of an investigational drug (not including investigational use of an approved drug) in the 30 days before the first dose of rhMBL.
* Prior liver transplants.
* Systemic chemotherapy within 1 year before liver transplantation.
* Serum creatinine >5 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of rhMBL administered i.v. at doses of 0.5 and 1.0 mg/kg, as 8 weekly doses over 8 weeks, in the setting of liver transplantation | 3 months

SECONDARY OUTCOMES:
Determine the pharmacokinetic (PK) profile of rhMBL | 3 months
Determine the pharmacodynamics (PD) (complement deposition) of rhMBL | 3 months
Determine the immunogenicity of rhMBL by testing for the presence of anti-rhMBL antibodies | 3 months
Detect preliminary evidence of activity of rhMBL by analyzing the incidence of infectious complications. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison Freifeld, MD, Principal Investigator — University of Nebraska Medical Center, 985400 Nebraska Medical Center, Omaha, NE 68198-5400
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai School of Medicine, New York, New York
  - Vanderbilt University, Nashville, Tennessee